CLINICAL TRIAL: NCT05833750
Title: Investigation of the Effect of Reflexology on Fatigue Parameter in Renal Transplantation Patients
Brief Title: Effects of Reflexology in Transplant Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sanko University (Other)
Responsible Party: Principal Investigator, hatıceguzel, directör, Sanko University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: haticeguzel
Record Dates: First submitted 2023-03-27; First posted 2023-04-27 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Renal Transplantation; Reflexology; Fatigue; Nursing
MeSH Terms: conditions — Fatigue | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Participant
Masking Description: participants'personal information is hidden
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- reflexology (Active Comparator): Patients in the reflexology group were applied twice a week for eight weeks.
  Interventions: Other: Reflexology
- Control group (No Intervention): No intervention was made

INTERVENTIONS:
Other: Reflexology — In the intervention group, reflexology was applied to the feet twice a week for 8 weeks.
  Arms: reflexology

SUMMARY:
Abstract Objective: The aim of this study is to examine the effect of reflexology on fatigue in kidney transplant patients.

Design: The study will be conducted as randomized, controlled and experimental. Method: The data of the research will be collected in the transplant clinic of a foundation university practice and research hospital between 07.12.2020 - 18.06.2021.

While the population of the study consisted of 254 patients who underwent kidney transplantation in the transplant unit, 68 patients were included in the sample. The patients included in the study were divided into reflexology (n=34) and control (n=34) groups with the help of a program. Data will be collected using Questionnaire and Piper Fatigue Scale. Chi-square test, Student's t test, Mann Whitney U test and Kruskal-Wallis test, correlation, generalized estimation equation and Least Significant Difference tests will be used in the evaluation of the data.

Keywords: kidney transplantation, reflexology, fatigue, nursing.

DETAILED DESCRIPTION:
Chronic kidney failure (CKD), the incidence of which continues to increase day by day and causes serious health problems in Turkey as in the world, maintains its current status as an important health problem. In the Chronic Kidney Diseases Prevalence (CREDIT) study in Turkey conducted by the Turkish Society of Nephrology (TSN), the incidence of CRF was found to be 15.7%, and the incidence of advanced stage CRF was 5.2%. As it is known, when this health problem reaches the stage of end-stage renal disease (ESRF), one of the renal replacement therapies (RRT) is absolutely needed.

Among the commonly used RRTs today are hemodialysis (HD), peritoneal dialysis (PD) and kidney transplantation (RTx). It has been reported that the best treatment option in terms of quality of life and patient survival is RTx. This is because a successful RTx significantly reduces the risk of mortality and morbidity compared to dialysis. According to the 2020 data of the Ministry of Health, HD was applied to 72.66% of the patients who received RRT, PD to 4.06% and RTx to 23.28%. According to the National Nephrology, Dialysis and Transplant Registration System Report, the number of RTx from live donors in Turkey in 2020 is 2,250 (90.04%), the number of RTx from cadavers is 249 (9.96%), this number is 2,499 in total.

2. BACKGROUND It is known that patients with ESRD likely experience a range of symptoms including nausea, vomiting, pain and fatigue. Therefore, patients prefer RTx more to stop dialysis and maintain a normal life. However, it is stated in the literature that fatigue continues after RTx. Fatigue is a subjective problem that affects individuals physically and psychologically and impairs their quality of life. For this reason, it is very important for nurses who are in constant communication with the patient to evaluate this symptom and to plan and implement appropriate nursing interventions. In this respect, it is recommended to use evidence-based approaches in the prevention and management of fatigue, to repeat the personalized training program at certain intervals, and to use integrative methods that can facilitate coping with fatigue. Exercise, yoga, acupressure and reflexology are among the most preferred integrative methods today. Different studies have reported that patients benefit from reflexology to reduce fatigue.

Reflexology is the method of applying physical pressure to all body parts, organs and reflex points corresponding to the endocrine glands in the ears, hands and feet, which are accepted as the mirror of the body, using certain finger and hand techniques. It has been reported that this approach facilitates relaxation, releases endorphins, modulates pain transmission and pain perception, regulates blood circulation and hemodynamic variables, and improves sleep quality. However, when the literature is examined, it has been seen that there are a limited number of studies evaluating the effect of reflexology in the management of fatigue after RTx. For this reason, this study was conducted to evaluate the effect of reflexology applied to patients who underwent RTx on fatigue, to contribute to fatigue management and to form a basis for future research.

3 STUDY 3.1 Purpose This study will be conducted to examine the effect of reflexology applied to kidney transplant patients on fatigue.

The Hypothesis of the Study Hypothesis -0 (H0): Reflexology applied to renal transplant patients does not reduce fatigue.

Hypothesis -1 (H1): Reflexology applied to renal transplant patients reduces fatigue.

3.2 Design The data of this randomized, controlled and experimental study will be obtained from patients admitted to the Organ Transplant Clinic of a Foundation University Hospital. Power analysis will be used to determine the sample size of the study.

3.3 Participants The population of the study consisted of 254 patients who underwent RTx in the Organ Transplant Unit. According to the power analysis, with the medium effect size (dz=0.5) and the minimum sample size required for the before-after comparison, it was planned to include a total of 68 patients, 34 per group, and the study will be completed with 68 patients. After the pre-test data of 68 patients who accepted to participate in the study were collected by the researcher, two groups will be randomly created by randomization method in the computer program based on the Piper Fatigue Scale (PFS) total scores. After the first patient is selected to one of the groups, the second patient will be automatically assigned to the second group. Assignment will continue until the blocks in each group are equal. Patients who volunteered to participate in the study, aged 18-75, had a kidney transplant, had a PFS score of 1 and above, had no communication problems, had a kidney transplant and were discharged from the hospital for at least 3 months. residing in the province where the research was conducted, will be included in the study. Patients who scored 0 on PFS, had open foot wounds, fractures, burns, and suspected thrombocytopenia, were diagnosed with deep vein thrombosis and peripheral neuropathy by the physician, and did not volunteer to participate in the study will be excluded from the study. The application will continue by assigning new patients to replace the withdrawn patients. Data collection tools will be applied after the patients included in the study are informed about the purpose of the study and the application stages. Participants in both patient groups will have informed consent forms signed.

3.4.1 Application of Data Collection Tools The researcher and the responsible physician of the relevant clinic received certification training in reflexology before the study. PFS will be applied to patients in both groups. As a result of the literature review, a total of 16 sessions of reflexology lasting 30 minutes each will be applied twice a week for eight weeks. At the end of the first month and the second month, PFS will be applied again to the patients in both groups. In addition, a session of reflexology will be applied to the patients in the control group after PFS is applied for the third time.

3.4.2 Reflexology Practice The patient will be taken to a single room with a bathroom in the transport unit for reflexology practice, considering his own privacy. The patient will lie on the bed after washing his feet in the bathroom and drying them with a paper towel. He will be placed in a semi-winged or supine position supporting his neck, waist and knees. The practitioner will wash their hands and rub them with some vaseline so that they have body temperature. He will then start reflexology with his right foot and continue to practice with his left foot. He will do the following methods for five minutes to warm his feet; Rotation and stretching of the Achilles tendon, bilateral ankle relaxation, and swelling from heel to toes and then from top of foot to ankle. During the application, the pressure with one hand will be supported by the other hand and both hands will be used actively.

Then, the pituitary, thyroid, parathyroid and adrenal glands and solar plexus points will be stimulated for 5 minutes to assess fatigue. Each pressure was applied for about 5-10 seconds and will be repeated 5-10 times. In the final stage, stretching the Achilles tendon, applying pressure to the solar plexus and effleurage movements will be applied for five minutes. While taking a deep breath, the patient's solar plexus will be pressed lightly, he will be asked to hold his breath during the pressure, and the process will be terminated by reducing the pressure applied to the point while exhaling. Then the same steps will be applied for the left foot. Thus, reflexology will be applied to both feet for a total of 30 minutes (15 minutes on each foot). After the procedure is completed, the patient will be allowed to rest for 5-10 minutes. During the application, the environment will be arranged as quiet and calm as possible so that the researcher and the patient can concentrate.

3.5 Ethical considerations Clinical Research Ethics Committee approval (2019/459/(Ver:2)) was obtained before starting the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients, who were voluntary to participate in the study, aged between 18-75 years,
* underwent renal transplantation,
* had a PFS score of 1 or higher,
* had no communication problem
* underwent renal transplantation and
* were discharged from the hospital for at least three months,
* were residing in the -province, where the study was conducted, were included in the study.

Exclusion Criteria:

* who got 0 point on PFS, had open foot wounds,
* suspected fractures,
* burns and thrombocytopenia, were diagnosed with deep vein thrombosis and peripheral --neuropathy by the physician
* were not voluntary to participate in the study, were excluded from the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-06-18 (Actual)

PRIMARY OUTCOMES:
Fatigue | 8 weeks
  Piper Fatigue Scale: Fatigue Scale VAS is between 0-10 points and consists of 22 items. It has four sub-dimensions. Total fatigue score is obtained by summing the items and dividing them by the total number of items. Score increase; indicates an increased level of fatigue

CONTACTS AND LOCATIONS:
Overall Officials: Hatice GUZEL, Study Director — Sanko University
Locations (1):
- Sanko university, Gaziantep, Şehitkamil, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No